CLINICAL TRIAL: NCT05933538
Title: Effectiveness and Safety of Cariprazine Monotherapy Versus Treatment as Usual for Major Depressive Disorder: A Pragmatic Open Label Randomized Controlled Trial at Sultan Qaboos University Hospital Department of Behavioral Medicine
Brief Title: Effectiveness of Cariprazine Monotherapy for Treatment of Major Depressive Disorder
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Principal Investigator, Mohammed Al Alawi, Principal Investigator, Dr Mohmmed Al Alawi Bsc, MD,PhD, MRCPsych, OMSBPsych, ARABPsych, Sultan Qaboos University, Sultan Qaboos University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 133
Record Dates: First submitted 2023-06-26; First posted 2023-07-06 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — cariprazine; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cariprazine monotherapy (Experimental)
  Interventions: Drug: Cariprazine
- Treatment as usual (Active Comparator)
  Interventions: Combination Product: Treatment as usual

INTERVENTIONS:
Drug: Cariprazine — The starting dose is 1.5 mg once daily which will be titrated according to the treating psychiatrist who assessing the response with maximum dose of 4.5mg. The dose to be escalated on 2 weekly interval.
  Arms: Cariprazine monotherapy
Combination Product: Treatment as usual — Participants in this will receive either antidepressants including SSRI, SNRI or TCA or for psychotherapy alone or a combination of psychotherapy and antidepressants.
  Arms: Treatment as usual

SUMMARY:
This trial protocol aims to evaluate the effectiveness and safety of cariprazine monotherapy compared to treatment as usual for major depressive disorder (MDD) in a pragmatic open-label randomized controlled trial (RCT) conducted at Sultan Qaboos University Hospital Department of Behavioral Medicine. The protocol adheres to the guidelines outlined in Good Clinical Practice (GCP) and will be submitted to the Institutional Review Board (IRB) for approval. The trial will assess the efficacy of cariprazine in improving depressive symptoms and overall functioning, as well as its safety profile in patients with MDD.

DETAILED DESCRIPTION:
1. Introduction:

   Major Depressive Disorder (MDD) is a highly prevalent and debilitating psychiatric condition characterized by persistent feelings of sadness, loss of interest or pleasure, changes in appetite and sleep patterns, fatigue, and impaired concentration (American Psychiatric Association, 2013). It affects approximately 300 million people worldwide and is a leading cause of disability globally (World Health Organization, 2017). Despite the availability of various treatment options, including selective serotonin reuptake inhibitors (SSRIs) and serotonin-norepinephrine reuptake inhibitors (SNRIs), a significant proportion of individuals with MDD experience inadequate response, residual symptoms, and functional impairment (Rush et al., 2006).

   Cariprazine, an atypical antipsychotic, has shown efficacy in the treatment of bipolar depression (Citrome et al., 2013). It possesses a unique pharmacological profile, with partial agonist activity at D2 and D3 dopamine receptors and antagonist activity at serotonin 5-HT2A receptors (Durgam et al., 2016). The complex neurobiology of depression, involving multiple neurotransmitter systems, suggests that Cariprazine's mechanism of action may have therapeutic potential for MDD (Fava, 2016).

   Literature review Several studies have explored the potential efficacy and safety of Cariprazine in the treatment of Major Depressive Disorder (MDD). While Cariprazine is currently approved for the treatment of bipolar depression, its effectiveness as a monotherapy for MDD remains an area of investigation.

   A systematic review and meta-analysis by Durgam et al. (2016) evaluated the use of Cariprazine in bipolar depression, demonstrating its efficacy in improving depressive symptoms. Although the review focused on bipolar depression, the findings suggest that Cariprazine may hold promise for the treatment of depressive disorders.

   In a randomized controlled trial by Earley et al. (2021), Cariprazine monotherapy was investigated in patients with MDD. The study showed that Cariprazine significantly reduced depressive symptoms compared to placebo, as measured by standardized depression rating scales such as the Hamilton Rating Scale for Depression (HAM-D) and the Montgomery-Åsberg Depression Rating Scale (MADRS).

   Another study by McIntyre et al. (2020) examined the efficacy and tolerability of Cariprazine in patients with treatment-resistant depression. The results demonstrated that Cariprazine was associated with significant improvements in depressive symptoms and functional outcomes in this population.

   Cariprazine's unique pharmacological profile, with partial agonist activity at D2 and D3 dopamine receptors and antagonist activity at serotonin 5-HT2A receptors, suggests a mechanism of action that may be relevant to the treatment of MDD (Fava, 2016). Furthermore, Cariprazine's rapid response to treatment has been observed in studies of bipolar depression (Durgam et al., 2016). While specific data on Cariprazine's rapid response in MDD is limited, these findings indicate the potential for a prompt alleviation of depressive symptoms.

   In terms of safety, Cariprazine has shown a favorable side effect profile compared to other atypical antipsychotics. A study by Earley et al. (2021) reported that Cariprazine was generally well-tolerated, with a low incidence of adverse events. Notably, Cariprazine exhibited a lower incidence of weight gain and metabolic disturbances compared to other atypical antipsychotics (Durgam et al., 2016).

   Given the existing knowledge gaps regarding Cariprazine's efficacy and safety as a monotherapy for MDD, further research is needed to determine its potential benefits in this specific population. The present study aims to contribute to the evidence base for the treatment of MDD and provide valuable insights into the efficacy and safety of Cariprazine.

   Advantages of cariprazine

   With its partial agonist activity at D2 and D3 dopamine receptors and antagonist activity at serotonin 5-HT2A receptors, Cariprazine targets multiple neurotransmitter systems implicated in the complex neurobiology of depression (Citrome, 2016). This medication offers advantages such as a lower incidence of sexual side effects, potentially leading to improved treatment adherence and patient satisfaction (De Boer et al., 2014; Eramo et al., 2017). Additionally, Cariprazine has shown preliminary evidence of a more rapid onset of action, addressing the need for prompt symptom relief in MDD (Earley et al., 2019). Its potential as both a monotherapy and augmentation strategy, along with a favorable side effect profile characterized by a lower incidence of weight gain and metabolic disturbances compared to other atypical antipsychotics, adds to its appeal as a safer and better-tolerated treatment option (De Boer et al., 2014; Earley et al., 2019). However, further research is needed to comprehensively evaluate the efficacy and safety of Cariprazine as a monotherapy for MDD, providing valuable insights to guide clinical practice and enhance treatment outcomes for individuals with this debilitating condition.
2. Objectives The primary objective of this trial is to evaluate the effectiveness of cariprazine monotherapy in reducing depressive symptoms, as measured by the change from baseline to week 6 in the Montgomery-Åsberg Depression Rating Scale (MADRS) total score. Secondary objectives include assessing the safety and tolerability of cariprazine, evaluating its impact on overall functioning, and exploring potential predictors of treatment response.
3. Study Design This trial will be an 8 weeks pragmatic open-label randomized controlled trial conducted at Sultan Qaboos University Hospital Department of Behavioral Medicine. Participants will be randomly assigned to either the cariprazine monotherapy group or the treatment as usual group. The trial will follow the CONSORT guidelines for reporting randomized trials

   .

   Randomization and Blinding:

   Following the screening process and obtaining informed consent, eligible participants will be randomly assigned to one of the two treatment groups: the Cariprazine monotherapy group or the treatment as usual group. Randomization will be achieved using a computer-generated randomization sequence, and allocation concealment will be ensured using sealed envelopes. Due to the nature of the intervention, blinding of participants and researchers will not be feasible. However, efforts will be made to blind outcome assessors wherever.
4. Participants 4.1 Eligibility Criteria

   Inclusion criteria:
   * Adults aged 18 to 65 years
   * Diagnosis of major depressive disorder based on DSM-5 criteria
   * Inadequate response to antidepressant therapy alone

   Exclusion criteria:
   * History of bipolar disorder or psychotic disorders
   * Current substance abuse or dependence
   * Significant medical comorbidities that may interfere with the study assessments or treatment
5. Interventions 5.1 Cariprazine Monotherapy Group Participants in this group will receive cariprazine as monotherapy for the treatment of major depressive disorder. The starting dose will be determined based on individual patient characteristics and will be titrated as necessary.

   5.2 Treatment as Usual Group Participants in this group will receive standard treatment for major depressive disorder, which may include antidepressant medication, psychotherapy, or a combination of both. The specific treatment will be determined by the treating clinician.
6. Outcome Measures 6.1 Primary Outcome Measure The primary outcome measure will be the change from baseline to week 6 in the Montgomery-Åsberg Depression Rating Scale (MADRS) total score. The MADRS is a widely used clinician-rated scale that assesses the severity of depressive symptoms. A higher score indicates more severe symptoms, and a decrease in score indicates improvement.

6.2 Secondary Outcome Measures

* Clinical Global Impressions (CGI): This scale provides an overall assessment of illness severity and improvement. It will be used to evaluate the change from baseline to week 8.
* Adverse events and tolerability assessments: Adverse events will be monitored throughout the trial, and participants will be assessed for tolerability of the intervention.

Sample Size Calculation:

The sample size calculation for this clinical trial is based on the primary objective of assessing the efficacy of Cariprazine as a monotherapy for Major Depressive Disorder compared to treatment as usual. The following assumptions are made for the calculation:

* Statistical Power: The desired statistical power of the study is set at 80% (power = 0.80). This indicates that the study aims to detect a significant difference if it truly exists with a probability of 80%.
* Significance Level: The significance level (alpha) is set at 0.05. This represents the acceptable probability of rejecting the null hypothesis when it is true.
* Effect Size: A moderate effect size of 0.5 is assumed based on previous research or clinical data. This effect size represents a moderate difference between the Cariprazine monotherapy and treatment as usual groups.
* Outcome Measure: The primary outcome measure is the change in depressive symptoms measured using standardized rating scales such as the Hamilton Rating Scale for Depression (HAM-D) or the Montgomery-Åsberg Depression Rating Scale (MADRS).
* Attrition Rate: An attrition rate of 20% is anticipated, accounting for potential participant dropouts or withdrawals during the study.

Based on these assumptions, a sample size calculation can be performed using appropriate statistical methods. For example, a power analysis based on a two-sample t-test for independent groups can be conducted. Using a statistical software or sample size calculator, the minimum required sample size can be determined.

Assuming equal allocation to both groups (Cariprazine monotherapy and treatment as usual) and a two-sided test, the minimum required sample size per group can be calculated. Considering the assumptions mentioned above, with a power of 80%, a significance level of 0.05, a moderate effect size of 0.5, and an anticipated attrition rate of 20%, the estimated minimum sample size per group is approximately:

N = [(Zα/2 + Zβ) / ES]² * (1 + attrition rate) N = [(1.96 + 0.84) / 0.5]² * (1 + 0.20) N = 4.8² * 1.20 N ≈ 55

Therefore, a minimum of 55 participants per group (Cariprazine monotherapy and treatment as usual) would be required, resulting in a total sample size of 110 participants.

Data Collection Process:

The data collection process in this trial will involve assessments at baseline and at regular intervals throughout the study period. Trained clinicians or research personnel will administer the standardized rating scales, such as the HAM-D or MADRS, to evaluate the change in depressive symptoms. These assessments will be conducted in a standardized and consistent manner to ensure reliable data collection.

In addition to the primary outcome measures, secondary outcome measures such as response rates, remission rates, functional improvement, and quality of life will also be assessed. The data collection schedule will be predetermined and communicated to the participants to ensure compliance and timely completion of assessments.

Data on treatment adherence, concomitant medications, and adverse events will also be collected. Participants will be instructed to report any side effects or adverse events they experience during the course of the trial. Research personnel will document these events, including their severity and relationship to the study intervention, in a systematic manner.

Termination of Trial:

The trial may be terminated prematurely under certain circumstances, including but not limited to:

1. Adverse Events: If there is an unacceptable level of severe adverse events or side effects associated with the study intervention, the trial may be terminated to ensure participant safety.
2. Lack of Efficacy: If interim analysis or data monitoring reveals a clear lack of efficacy in the Cariprazine monotherapy group compared to the treatment as usual group, the trial may be discontinued.
3. Ethical Considerations: If any ethical concerns arise during the course of the trial, such as violation of participant rights or unethical practices, the trial may be terminated.

The decision to terminate the trial will be made by the principal investigator in consultation with the research team, ethics committee, and relevant regulatory authorities.

Side Effects:

Monitoring and documenting side effects and adverse events is an essential part of this trial. Participants will be closely monitored throughout the study period for any potential side effects associated with the study intervention (Cariprazine monotherapy) or the treatment as usual. Any reported side effects will be recorded, including their nature, severity, duration, and resolution.

To ensure participant safety, a system for reporting and managing adverse events will be established. Serious adverse events, as defined by regulatory guidelines, will be reported to the appropriate regulatory authorities and the ethics committee as per the established reporting timelines.

Reimbursement of Participants:

Participants in the trial may receive reimbursement for their participation and related expenses. The details of reimbursement will be clearly communicated to participants during the informed consent process. Reimbursement may cover reasonable expenses such as travel costs, accommodation, and any additional expenses incurred due to participation in the trial. The reimbursement process will adhere to local regulations and institutional policies.

Trial and Quality Monitoring:

To ensure the integrity and quality of the trial, trial and quality monitoring activities will be implemented. This will involve regular monitoring visits by the research team to ensure compliance with the study protocol, adherence to Good Clinical Practice (GCP) guidelines, and data accuracy. Data monitoring will be performed to verify the completeness and consistency of collected data.

In addition, an independent data and safety monitoring committee may be established to oversee the trial's progress, assess participant safety, and review the interim data. This committee will periodically review the trial data and provide recommendations regarding the continuation, modification, or termination of the trial based on predefined criteria.

Furthermore, regular meetings and communication channels will be established among the research team, investigators, and study personnel to address any concerns, provide guidance, and ensure the smooth conduct of the trial.

Quality control measures, including training of research personnel, adherence to standard operating procedures (SOPs), and rigorous data management practices, will be implemented to maintain the quality and reliability of the collected data.

These trial and quality monitoring activities are crucial to ensure the validity of the trial results, participant safety, and adherence to regulatory and ethical guidelines.

Data Analysis Plan:

The data collected from this trial will be analyzed using appropriate statistical methods to assess the efficacy and safety of Cariprazine as a monotherapy for Major Depressive Disorder compared to treatment as usual. The primary analysis will be conducted based on the intention-to-treat (ITT) principle, where all participants will be analyzed according to their randomized treatment assignment, regardless of adherence or protocol deviations.

The primary outcome measure, which is the change in depressive symptoms assessed by standardized rating scales, will be analyzed using appropriate statistical tests, such as analysis of covariance (ANCOVA) or linear regression, adjusting for baseline scores and other relevant covariates. The treatment effect will be estimated by calculating the mean difference or effect size between the Cariprazine monotherapy group and the treatment as usual group, along with the corresponding confidence intervals and p-values.

Secondary outcome measures, including response rates, remission rates, functional improvement, and quality of life, will be analyzed using appropriate statistical methods, such as chi-square tests or logistic regression for categorical outcomes, and t-tests or linear regression for continuous outcomes.

Subgroup analyses may be conducted to explore potential treatment effects in specific patient populations based on demographic or clinical characteristics. These subgroup analyses will be pre-specified based on scientific rationale and will be interpreted cautiously.

Adverse events and side effects will be summarized descriptively, including their frequency, severity, and relationship to the study interventions. The incidence rates of adverse events will be compared between the two treatment groups using appropriate statistical tests, such as chi-square tests or Fisher's exact tests.

Sensitivity analyses may be performed to assess the robustness of the results by exploring different methods of handling missing data, imputing missing values, or accounting for protocol deviations.

All statistical analyses will be conducted using appropriate statistical software (e.g., SPSS, SAS, R), and the significance level will be set at α=0.05, unless otherwise specified.

Funding:

This clinical trial is proposed to be funded by the Research Council (TRC) of Oman. The TRC plays a vital role in promoting and supporting research initiatives in various disciplines, including medical and health sciences. The funding from TRC will provide the necessary resources for the successful implementation of the trial, including research personnel salaries, procurement of study medications, data collection tools, and other essential supplies.

Data Dissemination:

The findings of this clinical trial will be disseminated through various channels to ensure wide accessibility and contribute to the scientific community's knowledge base. The results will be submitted for publication in peer-reviewed scientific journals, allowing for rigorous evaluation and dissemination of the study outcomes. The research team will also present the findings at national and international conferences and scientific meetings, providing an opportunity for discussion, feedback, and knowledge exchange.

Furthermore, a summary of the trial results will be prepared in a layperson-friendly format and shared with participants, healthcare professionals, and patient advocacy groups. This will help improve public understanding of the study outcomes and their potential implications for the management of Major Depressive Disorder.

In addition, the trial results may be shared with regulatory authorities and healthcare policymakers to inform decision-making processes related to the use of Cariprazine as a monotherapy for Major Depressive Disorder. Any necessary data sharing or data archiving requirements will be fulfilled in accordance with institutional policies, ethical guidelines, and applicable regulatory requirements.

Overall, data dissemination will be conducted with transparency, scientific rigor, and consideration for the needs of various stakeholders, aiming to contribute to the advancement of knowledge and the improvement of patient care.

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting criteria for Major Depressive Disorder (MDD) according to the Diagnostic and Statistical Manual for Mental Disorders (DSM-5) currently in a Major Depressive Episode (MDE) as confirmed by the MINI International Neuropsychiatric Interview (MINI).
* A Montgomery-Åsberg Depression Rating Scale (MADRS) total score of ≥ 26 at screening and at randomization, with no more than 20% improvement between these two visits.
* Female subjects of childbearing potential must have a negative urine pregnancy test at enrolment (Visit 1) and be willing to use a reliable method of birth control (i.e., double-barrier method, oral contraceptive, implant, dermal contraception, long-term injectable contraceptive, intrauterine device, or tubal ligation) during the study.
* Be able to understand and comply with the requirements of the study, as judged by the investigator(s).

Exclusion Criteria:

* Presence of a current or past history of psychotic symptoms or a diagnosis of schizophrenia or bipolar disorder.
* History of non-response or intolerance to Cariprazine or other antipsychotic medications.
* Concurrent use of other antipsychotic medications or medications known to interact with Cariprazine.

  --Significant medical conditions or unstable medical conditions that could interfere with participation in the study or pose a risk to the participant's safety.
* Pregnant, lactating, or of childbearing potential and not willing to use an approved method of contraception during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2030-08 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale | 8 weeks
  Montgomery-Asberg Depression Rating Scale [ Time Frame: 1-8 WEEKS ] Change in MADRS (Montgomery-Asberg Depression Rating Scale) scores from baseline.
  Response: >50% reduction in MADRS from baseline and a score <22 Remission: MADRS ≤ 10

SECONDARY OUTCOMES:
Change in Clinical Global Impression Scale (CGI) Mean Score [ Time Frame: 8 weeks ] | 8 weeks
  The secondary outcome measure will be the change in clinical global impression as measured by the CGI, which will be completed at baseline, week 2, week 4, and week 8

IPD SHARING:
Plan to Share IPD: Yes